CLINICAL TRIAL: NCT05280756
Title: Home-based Transcranial Direct-current Stimulation (tDCS) for Prevention of Suicidal Ideation
Brief Title: Home-based tDCS for Prevention of Suicidal Ideation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Brain & Behavior Research Foundation (Other)
Responsible Party: Principal Investigator, Yeates Conwell, MD, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: STUDY00008028
Record Dates: First submitted 2022-03-04; First posted 2022-03-15 (Actual); Results first posted 2025-05-07 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Suicidal Ideation
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active home-based transcranial direct current stimulation (tDCS) (Experimental): The active home-based tDCS delivers a constant current intensity of 2mA on the subject's scalp, with electrodes positioned bilaterally (anodal-left and cathodal-right), on the dorsolateral prefrontal cortex (DLPFC), for 30 minutes.
  Interventions: Device: Home-based transcranial direct current stimulation (tDCS)
- Sham home-based transcranial direct current stimulation (tDCS) (Sham Comparator): The sham home-based tDCS looks identical to a typical active home-based tDCS cap but delivers a 30-second ramp-up (0-2 mA) stimulation followed by a 30-second ramp-down (2-0 mA) at the beginning and end of the application.
  Interventions: Device: Sham home-based transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: Home-based transcranial direct current stimulation (tDCS) — Each participant will be asked to do ten home-based tDCS sessions, one per weekday, during two weeks (Monday to Friday). Each session will be supervised remotely by a member of the research staff via HIPAA-compliant videoconference. Participants will receive active home-based tDCS (constant current intensity of 2mA) anodal-left and cathodal-right prefrontal for 30 minutes per session daily for 2 weeks (Monday to Friday - 10 sessions overall) via a tDCS stimulator with headgear and 5x7 (35cm2) saline-soaked surface sponge electrodes.
  Other Names: Soterix 1X1 mini-CT Transcranial Direct Current Stimulation (tcDCS) device
  Arms: Active home-based transcranial direct current stimulation (tDCS)
Device: Sham home-based transcranial direct current stimulation (tDCS) — Each participant will be asked to do ten home-based sessions, one per weekday, during two weeks (Monday to Friday). Each session will be supervised remotely by a member of the research staff via HIPAA-compliant videoconference. Participants will receive sham home-based tDCS for 30 minutes per session daily for 2 weeks (Monday to Friday - 10 sessions overall) via a tDCS stimulator with headgear and 5x7 (35cm2) saline-soaked surface sponge electrodes.
  Other Names: Soterix 1X1 mini-CT Transcranial Direct Current Stimulation (tcDCS) device
  Arms: Sham home-based transcranial direct current stimulation (tDCS)

SUMMARY:
Risk for suicide is elevated in the period after discharge from hospital among adults with major affective disorder. The primary objective of this study is to investigate the feasibility of delivering tDCS sessions for high-risk patients for suicide at home in the days following discharge from an emergency department or inpatient unit. This is a single-center, randomized, sham-controlled, double-blind clinical study. We plan to assess up to 80 adult patients for eligibility over 12 months of which 20 will be enrolled and randomized. Clinical assessments will be performed at baseline, post-treatment day 14 (14 days after the first tDCS session), and follow-up day 30 and 60 (30 and 60 days after the first tDCS session, respectively).

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65 years
* diagnosis of mood or bipolar disorder registered in the electronic hospital medical record
* history of suicidal ideation and/or suicidal behavior at the time of admission registered in the electronic hospital medical record
* absent of suicidal ideation at the time of enrollment (defined as questions 1 and 2 of the C-SSRS answered "no")
* ability and willingness to provide information and permission to contact at least one person in the case of a need to contact them to promote subject safety or inability to reach the subject for follow-up
* a living situation with access to a private space suitable for the administration of the RS-tDCS sessions in the next three weeks
* agree to use a medically acceptable form of birth control while receiving the treatment if you are an individual able to become pregnant
* living in Monroe County region, as this is the area covered by the Mobile Crisis Team, a URMC psychiatric emergency team serving anyone within Monroe County
* device or computer with internet access for a URMC-approved remote RS-tDCS supervision
* ability to manage proper use of the device in a practice session

Exclusion Criteria:

* acute psychiatric instability or substance abuse (e.g., psychotic symptoms, alcohol misuse in the previous three months, use of any illicit drugs in the previous three months)
* unstable medical condition with reduction of functional capacity
* history of epilepsy or seizures in the last year
* history of neurodegenerative diseases registered in the electronic hospital medical record
* presence of or implanted any ferromagnetic metal in the head or the neck
* pregnant or breastfeeding or willingness to become pregnant in the next month
* history of head trauma (e.g., head injury, brain injury) or neurosurgery
* history of skin disorder or sensitive skin area near stimulation locations
* the presence of pacemaker
* current treatment with electroconvulsive therapy or transcranial magnetic stimulation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-09-21 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yeates Conwell, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
We are investigating options for making unidentifiable research data from individual participants available for public sources such as Harvard Dataverse.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Excluded (n=24) Not meeting inclusion criteria (n=11) Declined to participate (n=3) Refused questioning (n=1) Exclusion criteria (n=5) Unable to approach (n=4)
Period: Overall Study
Arm/Group | Active Home-based Transcranial Direct Current Stimulation (tDCS) | Sham Home-based Transcranial Direct Current Stimulation (tDCS)
Started | 5 | 4
Completed | 4 | 3
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Home-based Transcranial Direct Current Stimulation (tDCS) | Sham Home-based Transcranial Direct Current Stimulation (tDCS) | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.80 (2.68) | 22.00 (2.45) | 21.89 (2.42)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Male | 1 | 0 | 1
  Sex: Female | 2 | 3 | 5
  Sex: Transgender (Male-to-Female) | 1 | 0 | 1
  Sex: Transgender (Female-to-Male) | 1 | 0 | 1
  Sex: Not sure (non-binary) | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White/Non-Hispanic | 5 | 2 | 7
  Race: Hispanic or Latino | 0 | 1 | 1
  Race: Black or African American | 0 | 1 | 1
History of suicidal ideation or behavior at hospital admission [Count of Participants; unit: Participants] | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of the Intervention: Number of Participants Who Completed 5 or More Remotely Supervised Transcranial Direct Current Stimulation (RS-tDCS) Sessions
Description: Number of completed remotely supervised transcranial direct current stimulation (RS-tDCS) sessions, for both active and sham groups: We expect at least 70% of the subjects to complete at least 5 of recommended 10 RS-tDCS sessions.
Time Frame: 14 days after start of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Active Home-based Transcranial Direct Current Stimulation (tDCS) | Sham Home-based Transcranial Direct Current Stimulation (tDCS)
Number analyzed (Participants) | 5 | 4
Participants | 4 | 3

2. Secondary Outcome: Mean Intensity of Suicidal Ideation as Assessed by the Columbia Suicide Severity Rating Scale (C-SSRS) Day 14
Description: The C-SSRS (Columbia-Suicide Severity Rating Scale) is a suicidal ideation and behavior rating scale. For the 5 items assessing suicidal ideation intensity, each item is scored 0-5. The total intensity score is the sum of these 5 items (range 0-25), with higher scores indicating greater suicidal ideation. The mean is calculated by the sum of the scores of the participants at Day 14 divided by the number of participants
Time Frame: day 14 [+ 7 days] from the first RS-tDCS session
Population: All participants who completed both baseline and Day 14 C-SSRS assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Home-based Transcranial Direct Current Stimulation (tDCS) | Sham Home-based Transcranial Direct Current Stimulation (tDCS)
Number analyzed (Participants) | 4 | 3
score on a scale | 8.25 (10.53) | 6.33 (10.97)

3. Secondary Outcome: Mean Intensity of Suicidal Ideation as Assessed by the Columbia Suicide Severity Rating Scale (C-SSRS) Day 30
Description: The C-SSRS (Columbia-Suicide Severity Rating Scale) is a suicidal ideation and behavior rating scale. For the 5 items assessing suicidal ideation intensity, each item is scored 0-5. The total intensity score is the sum of these 5 items (range 0-25), with higher scores indicating greater suicidal ideation. The mean is calculated by the sum of the scores of the participants at Day 30 divided by the number of participants
Time Frame: Day 30 (± 7 days) from the first RS-tDCS session
Population: All participants who completed both baseline and Day 30 C-SSRS assessments were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Home-based Transcranial Direct Current Stimulation (tDCS) | Sham Home-based Transcranial Direct Current Stimulation (tDCS)
Number analyzed (Participants) | 4 | 3
score on a scale | 9.00 (10.52) | 7.33 (12.70)

4. Secondary Outcome: Mean Intensity of Suicidal Ideation as Assessed by the Columbia Suicide Severity Rating Scale (C-SSRS) Day 60
Description: Outcome measure description: The C-SSRS (Columbia-Suicide Severity Rating Scale) is a suicidal ideation and behavior rating scale. For the 5 items assessing suicidal ideation intensity, each item is scored 0-5. The total intensity score is the sum of these 5 items (range 0-25), with higher scores indicating greater suicidal ideation. The mean is calculated by the sum of the scores of the participants at Day 60 divided by the number of participants
Time Frame: Day 60 (± 10 days) from the first RS-tDCS session
Population: All participants who completed both baseline and Day 60 C-SSRS assessments were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Home-based Transcranial Direct Current Stimulation (tDCS) | Sham Home-based Transcranial Direct Current Stimulation (tDCS)
Number analyzed (Participants) | 4 | 3
score on a scale | 6.50 (7.89) | 10.00 (9.54)

5. Secondary Outcome: Acceptability of the Intervention as Assessed by Participant-reported Questionnaire
Description: Acceptability of the intervention is assessed based on participants' readiness, self-confidence, and satisfaction with treatment. Specifically, acceptability is determined if at least 60% of participants respond "Strongly agree" or "Agree" to item 11 of the acceptability questionnaire: "Overall, I felt that transcranial electrical stimulation treatment benefited me." The questionnaire uses a 5-point Likert scale: "Strongly agree," "Agree," "Neither agree nor disagree," "Disagree," "Strongly disagree." Higher scores indicate greater perceived acceptability.
Time Frame: Collected after the final RS-tDCS session (tenth session)
Population: All participants who completed the acceptability questionnaire after the final RS-tDCS session.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Home-based Transcranial Direct Current Stimulation (tDCS) | Sham Home-based Transcranial Direct Current Stimulation (tDCS)
Number analyzed (Participants) | 4 | 3
Participants | 2 | 1

6. Secondary Outcome: Proportion of Patients With no Suicidal Ideation as Assessed by the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: Proportion of participants who report no suicidal ideation, defined as answering "No" to both question 1 ("Have you wished you were dead or wished you could go to sleep and not wake up?") and question 2 ("Have you actually had any thoughts of killing yourself?") on the C-SSRS. Higher proportions indicate fewer participants experiencing suicidal ideation.
Time Frame: day 14 [+ 7 days] from the first RS-tDCS session
Population: All participants who completed both baseline and Day 14 C-SSRS assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Home-based Transcranial Direct Current Stimulation (tDCS) | Sham Home-based Transcranial Direct Current Stimulation (tDCS)
Number analyzed (Participants) | 4 | 3
Participants | 2 | 2

7. Secondary Outcome: Proportion of Patients With no Suicidal Ideation as Assessed by the C-SSRS
Description: as for outcome 6
Time Frame: day 30 [+ 7 days] from the first RS-tDCS session
Population: All participants who completed both baseline and Day 30 C-SSRS assessments
Measure: Count of Participants; unit: Participants
Arm/Group | Active Home-based Transcranial Direct Current Stimulation (tDCS) | Sham Home-based Transcranial Direct Current Stimulation (tDCS)
Number analyzed (Participants) | 4 | 3
Participants | 2 | 2

8. Secondary Outcome: Proportion of Patients With no Suicidal Ideation as Assessed by the C-SSRS
Description: as for outcome 6
Time Frame: day 60 [+ 10 days] from the first RS-tDCS session
Population: All participants who completed both baseline and Day 60 C-SSRS assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Home-based Transcranial Direct Current Stimulation (tDCS) | Sham Home-based Transcranial Direct Current Stimulation (tDCS)
Number analyzed (Participants) | 4 | 3
Participants | 1 | 1

9. Secondary Outcome: Mean Intensity of Rumination as Assessed by the Ruminative Responses Scale (RRS) Day 14
Description: The Ruminative Responses Scale (RRS) is a 22-item self-report measure assessing rumination. Each item is rated on a 4-point Likert scale: 1 = almost never, 2 = sometimes, 3 = often, 4 = almost always. The total score is calculated by summing the scores of all 22 items (range 22-88), with higher scores indicating greater rumination. The mean is calculated by the sum of the scores of the participants at Day 14 divided by the number of participants
Time Frame: day 14 [+ 7 days] from the first RS-tDCS session
Population: All participants who completed both baseline and Day 14 RRS assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Home-based Transcranial Direct Current Stimulation (tDCS) | Sham Home-based Transcranial Direct Current Stimulation (tDCS)
Number analyzed (Participants) | 4 | 3
score on a scale | 58.25 (12.04) | 63.33 (9.87)

10. Secondary Outcome: Mean Intensity of Rumination as Assessed by the Ruminative Responses Scale (RRS) Day 30
Description: The Ruminative Responses Scale (RRS) is a 22-item self-report measure assessing rumination. Each item is rated on a 4-point Likert scale: 1 = almost never, 2 = sometimes, 3 = often, 4 = almost always. The total score is calculated by summing the scores of all 22 items (range 22-88), with higher scores indicating greater rumination. The mean is calculated by the sum of the scores of the participants at Day 30 divided by the number of participants
Time Frame: day 30 [+ 7 days] from the first RS-tDCS session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Home-based Transcranial Direct Current Stimulation (tDCS) | Sham Home-based Transcranial Direct Current Stimulation (tDCS)
Number analyzed (Participants) | 4 | 3
score on a scale | 54 (17.15) | 52 (14.73)

11. Secondary Outcome: Mean Intensity of Rumination as Assessed by the Ruminative Responses Scale (RRS) Day 60
Description: The Ruminative Responses Scale (RRS) is a 22-item self-report measure assessing rumination. Each item is rated on a 4-point Likert scale: 1 = almost never, 2 = sometimes, 3 = often, 4 = almost always. The total score is calculated by summing the scores of all 22 items (range 22-88), with higher scores indicating greater rumination. The mean is calculated by the sum of the scores of the participants at Day 60 divided by the number of participants
Time Frame: day 60 [+ 10 days] from the first RS-tDCS session
Population: All participants who completed both baseline and Day 60 RRS assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Home-based Transcranial Direct Current Stimulation (tDCS) | Sham Home-based Transcranial Direct Current Stimulation (tDCS)
Number analyzed (Participants) | 4 | 3
score on a scale | 51 (20.17) | 55 (6.24)

12. Secondary Outcome: Mean Symptoms Associated With Suicidal Ideation as Assessed by the Concise Associated Symptoms Tracking (CAST) Scale Day 14
Description: The Concise Associated Symptoms Tracking (CAST) scale is a 16-item self-report measure assessing symptoms associated with suicidal ideation across five domains: anxiety (3 items, subscore range 3-15), irritability (5 items, subscore range 5-25), mania (4 items, subscore range 4-20), insomnia (2 items, subscore range 2-10), and panic (2 items, subscore range 2-10). Total CAST scores range from 16 to 80. Each item is rated on a 5-point Likert scale: 1 = strongly disagree, 2 = disagree, 3 = neither agree nor disagree, 4 = agree, 5 = strongly agree. Higher scores indicate greater symptom severity. The mean is calculated by the sum of the scores of the participants at Day 14 divided by the number of participants
Time Frame: day 14 [+ 7 days] from the first RS-tDCS session
Population: All participants who completed both baseline and Day 14 CAST assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Home-based Transcranial Direct Current Stimulation (tDCS) | Sham Home-based Transcranial Direct Current Stimulation (tDCS)
Number analyzed (Participants) | 4 | 3
score on a scale | 45.5 (9.98) | 47.33 (10.79)

13. Secondary Outcome: Mean Symptoms Associated With Suicidal Ideation as Assessed by the Concise Associated Symptoms Tracking (CAST) Scale Day 30
Description: The Concise Associated Symptoms Tracking (CAST) scale is a 16-item self-report measure assessing symptoms associated with suicidal ideation across five domains: anxiety (3 items, subscore range 3-15), irritability (5 items, subscore range 5-25), mania (4 items, subscore range 4-20), insomnia (2 items, subscore range 2-10), and panic (2 items, subscore range 2-10). Total CAST scores range from 16 to 80. Each item is rated on a 5-point Likert scale: 1 = strongly disagree, 2 = disagree, 3 = neither agree nor disagree, 4 = agree, 5 = strongly agree. Higher scores indicate greater symptom severity. The mean is calculated by the sum of the scores of the participants at Day 30 divided by the number of participants
Time Frame: day 30 [+ 7 days] from the first RS-tDCS session
Population: All participants who completed both baseline and Day 30 CAST assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Home-based Transcranial Direct Current Stimulation (tDCS) | Sham Home-based Transcranial Direct Current Stimulation (tDCS)
Number analyzed (Participants) | 4 | 3
score on a scale | 42.25 (2.63) | 46.67 (13.20)

14. Secondary Outcome: Mean Symptoms Associated With Suicidal Ideation as Assessed by the Concise Associated Symptoms Tracking (CAST) Scale Day 60
Description: The Concise Associated Symptoms Tracking (CAST) scale is a 16-item self-report measure assessing symptoms associated with suicidal ideation across five domains: anxiety (3 items, subscore range 3-15), irritability (5 items, subscore range 5-25), mania (4 items, subscore range 4-20), insomnia (2 items, subscore range 2-10), and panic (2 items, subscore range 2-10). Total CAST scores range from 16 to 80. Each item is rated on a 5-point Likert scale: 1 = strongly disagree, 2 = disagree, 3 = neither agree nor disagree, 4 = agree, 5 = strongly agree. Higher scores indicate greater symptom severity. The mean is calculated by the sum of the scores of the participants at Day 60 divided by the number of participants
Time Frame: day 60 [+ 10 days] from the first RS-tDCS session
Population: All participants who completed both baseline and Day 60 CAST assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Home-based Transcranial Direct Current Stimulation (tDCS) | Sham Home-based Transcranial Direct Current Stimulation (tDCS)
Number analyzed (Participants) | 4 | 3
score on a scale | 44.75 (12.53) | 45 (3.61)

15. Secondary Outcome: Mean Depression Severity as Assessed by the Montgomery-Asberg Depression Rating Scale (MADRS) Day 14
Description: MADRS is a 10-item clinician-administered questionnaire assessing the following symptoms: 1) Apparent sadness, 2) Reported sadness, 3) Inner tension, 4) Reduced sleep, 5) Reduced appetite, 6) Concentration difficulties, 7) Lassitude, 8) Inability to feel, 9) Pessimistic thoughts, 10) Suicidal thoughts. Each item is scored 0-6, giving a total score range of 0-60. Higher scores indicate more severe depressive symptoms. The mean is calculated by the sum of the scores of the participants at Day 14 divided by the number of participants
Time Frame: day 14 [+ 7 days] from the first RS-tDCS session
Population: All participants who completed both baseline and Day 14 MADRS assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Home-based Transcranial Direct Current Stimulation (tDCS) | Sham Home-based Transcranial Direct Current Stimulation (tDCS)
Number analyzed (Participants) | 4 | 3
score on a scale | 20.25 (19.05) | 30.67 (15.31)

16. Secondary Outcome: Mean Depression Severity as Assessed by the Montgomery-Asberg Depression Rating Scale (MADRS) Day 30
Description: MADRS is a 10-item clinician-administered questionnaire assessing the following symptoms: 1) Apparent sadness, 2) Reported sadness, 3) Inner tension, 4) Reduced sleep, 5) Reduced appetite, 6) Concentration difficulties, 7) Lassitude, 8) Inability to feel, 9) Pessimistic thoughts, 10) Suicidal thoughts. Each item is scored 0-6, giving a total score range of 0-60. Higher scores indicate more severe depressive symptoms. The mean is calculated by the sum of the scores of the participants at Day 30 divided by the number of participants
Time Frame: day 30 [+ 7 days] from the first RS-tDCS session
Population: All participants who completed both baseline and Day 30 MADRS assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Home-based Transcranial Direct Current Stimulation (tDCS) | Sham Home-based Transcranial Direct Current Stimulation (tDCS)
Number analyzed (Participants) | 4 | 3
score on a scale | 20.33 (20.26) | 25.33 (18.90)

17. Secondary Outcome: Mean Depression Severity as Assessed by the Montgomery-Asberg Depression Rating Scale (MADRS) Day 60
Description: MADRS is a 10-item clinician-administered questionnaire assessing the following symptoms: 1) Apparent sadness, 2) Reported sadness, 3) Inner tension, 4) Reduced sleep, 5) Reduced appetite, 6) Concentration difficulties, 7) Lassitude, 8) Inability to feel, 9) Pessimistic thoughts, 10) Suicidal thoughts. Each item is scored 0-6, giving a total score range of 0-60. Higher scores indicate more severe depressive symptoms. The mean is calculated by the sum of the scores of the participants at Day 60 divided by the number of participants
Time Frame: day 60 [+ 10 days] from the first RS-tDCS session
Population: All participants who completed both baseline and Day 60 MADRS assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Home-based Transcranial Direct Current Stimulation (tDCS) | Sham Home-based Transcranial Direct Current Stimulation (tDCS)
Number analyzed (Participants) | 4 | 3
score on a scale | 22 (18.13) | 18.67 (18.45)

18. Secondary Outcome: Mean Cumulative Side Effect Score Per Participant Across RS tDCS Sessions
Description: After each RS tDCS session (up to 10 sessions per participant), seven prespecified side effects itching, burning, headache, fatigue, nervousness, dizziness, and difficulty concentrating were assessed using the RS tDCS Side Effect Rating Scale. Each symptom was rated on a numeric scale from 0 to 10, where 0 indicates not at all and 10 indicates the highest degree of severity.
  For each participant and each symptom, ratings were summed across all completed sessions to generate a cumulative symptom specific side effect score, with a theoretical range of 0 to 100. Higher scores indicate greater cumulative side effect burden. Participants contributed all available session ratings with no imputation. For reporting, participant level cumulative scores were averaged across participants for each symptom and summarized as mean and standard deviation.
Time Frame: Assessed after each RS-tDCS session; values reported represent the average and summarized across all sessions completed during the 4-week treatment period
Population: All participants who completed the side effect questionnaire at the end of each RS tDCS session
Measure: Mean (Standard Deviation); unit: Score on a 0-100 scale
Arm/Group | Active Home-based Transcranial Direct Current Stimulation (tDCS) | Sham Home-based Transcranial Direct Current Stimulation (tDCS)
Number analyzed (Participants) | 4 | 3
Score on a 0-100 scale
  Itching | 14.00 (6.98) | 12 (17.44)
  Burning | 33.00 (16.69) | 13.33 (11.06)
  Headache | 13.25 (6.13) | 8.67 (10.97)
  Fatigue | 6.25 (3.95) | 1.33 (2.31)
  Nervousness | 2.50 (3.32) | 0.67 (1.16)
  Dizziness | 1.25 (1.89) | 0.00 (0.00)
  Difficult concentrating | 2.50 (3.11) | 3.00 (3.00)

19. Secondary Outcome: Number of Participants Reporting Solicited Side Effects During RS tDCS Treatment
Description: Predefined, expected side effects associated with RS tDCS were prospectively and systematically collected using a standardized post session side effect questionnaire administered after each RS tDCS session. Solicited side effects included itching, burning, headache, fatigue, nervousness, dizziness, difficulty concentrating, and other expected sensations related to stimulation.
  This outcome summarizes the number of participants who reported one or more solicited side effects at any time during the treatment period. These solicited side effect assessments were collected as part of structured safety monitoring and are reported as outcome measures rather than as adverse events. Unsolicited adverse events meeting ClinicalTrials.gov reporting criteria are reported separately in the Adverse Events module.
Time Frame: Assessed after each RS tDCS session during the 4 week treatment period
Population: All participants who completed at least one post session RS tDCS side effect questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Active Home-based Transcranial Direct Current Stimulation (tDCS) | Sham Home-based Transcranial Direct Current Stimulation (tDCS)
Number analyzed (Participants) | 4 | 3
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: 70 days
Arm/Group | Active Home-based Transcranial Direct Current Stimulation (tDCS) | Sham Home-based Transcranial Direct Current Stimulation (tDCS)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 2/5 | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Home-based Transcranial Direct Current Stimulation (tDCS) (N=5) | Sham Home-based Transcranial Direct Current Stimulation (tDCS) (N=4)
stress-related syncope (Nervous system disorders) | 1 (1) | 0 (0)
increased dose of SSRI (Psychiatric disorders) | 1 | 0 — The participant reported an SSRI dose adjustment since the prior assessment
Increased dose of SSRI (Psychiatric disorders) | 0 | 1 — The participant reported an SSRI dose adjustment since the prior assessment
decreased dose of SSRI (Psychiatric disorders) | 1 | 0 — The participant reported an SSRI dose adjustment since the prior assessment
discontinuation of NDRI (Psychiatric disorders) | 1 | 0 — The participant reported discontinuation of an NDRI since the prior assessment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-09): https://cdn.clinicaltrials.gov/large-docs/56/NCT05280756/Prot_SAP_001.pdf
  • Informed Consent Form (2023-10-09): https://cdn.clinicaltrials.gov/large-docs/56/NCT05280756/ICF_002.pdf